CLINICAL TRIAL: NCT04392388
Title: Health, Perception, Practices, Relations and Social Inequalities in the General Population During the Covid-19 Crisis - Serology
Brief Title: Health, Perception, Practices, Relations and Social Inequalities in the General Population During the Covid-19 Crisis
Acronym: SAPRIS-SERO
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C20-26; 2020-A01195-34 (Other: ID RCB (ANSM))
Record Dates: First submitted 2020-05-15; First posted 2020-05-18 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2024-02

CONDITIONS: SARS-CoV 2
Keywords: SARS-CoV2; cohort; containment; serology; prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serology samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SAPRIS-SERO: SAPRIS-SERO enrolls participants from cohorts entitled: Constances, E3N-E4N, ELFE, Epipage 2 and NutriNet-Santé.
  Interventions: Biological: Non applicable

INTERVENTIONS:
Biological: Non applicable — to collect data from questionnaires and to collect serological samples

SUMMARY:
This study aims to quantify and follow the cumulative incidence of SARS-CoV-2 infection in the French population using serological tests and to assess the determinants of infection from Constances, E3N-E4N, ELFE-Epipage 2 and NutriNet-Santé cohorts.

DETAILED DESCRIPTION:
The primary objective is to assess the cumulative incidence of infection in the general population using dried blood spot sampling.

The secondary objectives are:

* To identify factors associated with a positive SARS-CoV-2 infection (positive serology) and to characterize the durability of the serological response to SARS-CoV-2
* To identify associations of symptoms predictive of a SARS-CoV-2 infection
* To estimate the health care use associated with a SARS-CoV-2 infection
* To estimate the fraction of sub-clinical infections or infections not captured by the healthcare system;
* To study the acceptability of a mass anti-SARS-CoV-2 serological testing and the impact of its result, linked with social inequalities in health;
* To estimate the individual and collective impact of containment and other preventive measures on the risk of SARS-CoV-2 infection;
* To study the impact of social and territorial inequalities on seroprevalence levels.

ELIGIBILITY:
Inclusion Criteria:

* non applicable, already enrolled in the cohorts

Exclusion Criteria:

* non applicable

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants from cohorts entitled : Constances, E3N-E4N, ELFE, Epipage 2 and NutriNet-Santé
Sampling Method: Non-Probability Sample
Enrollment: 96883 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of SARS-Cov2 infection in the general population. | 8 months
  Simple and corrected estimate of the number of seropositive individuals/number of individuals at risk in different strata, based on weighting and calibration and taking into account the random cohort effect.

SECONDARY OUTCOMES:
Maintenance over time of the acquisition of anti-SARS-Cov2 antibodies | 8 months
  Decay kinetics estimated by mixed effect model with repeated data per subject
Rate of use of care (medical care, hospitalization, center 15) linked to the occurrence of symptoms suggestive of a SARS-Cov2 infection, and share attributable to the infection | 8 months
  Rate of use of care (medical care, hospitalization, center 15) linked to the occurrence of symptoms suggestive of a SARS-Cov2 infection, and share attributable to the infection during a time frame of 8 months
Proportion of infections without reported or pauci-symptomatic symptoms and their epidemiological and social determinants | 8 months
  Proportion of infections without reported or pauci-symptomatic symptoms and their epidemiological and social déterminants during a time frame of 8 months.
Proportion of tests proposed, accepted, performed, based on social and demographic characteristics | 8 months
  Proportion of tests proposed, accepted, performed, based on social and demographic characteristics during a time frame of 8 months.
Proportion and intensity of use of barrier measures (hydroalcoholic gel, mask, social distancing, description of outings / reasons, duration, frequency) and association with the level of seroprevalence | 8 months
  Proportion and intensity of use of barrier measures (hydroalcoholic gel, mask, social distancing, description of outings / reasons, duration, frequency) and association with the level of seroprevalence during a time frame of 8 months
Strengths of associations between socio-behavioral factors and level of seroprevalence | 8 months
  Strengths of associations between socio-behavioral factors and level of seroprevalence during a time frame of 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Carrat, MD, Principal Investigator — Inserm - Sorbonne Université
Locations (1):
- Inserm, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing is managed via the cohorts (Constances, E3N/E4N, NutriNetSante, Elfe/Epipage2) specific governing bodies.

REFERENCES:
- [Result] Robineau O, Zins M, Touvier M, Wiernik E, Lemogne C, de Lamballerie X, Blanche H, Deleuze JF, Saba Villarroel PM, Dorival C, Nicol J, Gomes-Rima R, Correia E, Coeuret-Pellicer M, Druesne-Pecollo N, Esseddik Y, Ribet C, Goldberg M, Severi G, Carrat F; Sante, Pratiques, Relations et Inegalites Sociales en Population Generale Pendant la Crise COVID-19-Serologie (SAPRIS-SERO) Study Group. Long-lasting Symptoms After an Acute COVID-19 Infection and Factors Associated With Their Resolution. JAMA Netw Open. 2022 Nov 1;5(11):e2240985. doi: 10.1001/jamanetworkopen.2022.40985. PMID 36350653
- [Result] Carrat F, Villarroel PMS, Lapidus N, Fourie T, Blanche H, Dorival C, Nicol J, Deleuze JF, Robineau O; SAPRIS-SERO Study Group; Touvier M, Severi G, Zins M, de Lamballerie X. Heterogeneous SARS-CoV-2 humoral response after COVID-19 vaccination and/or infection in the general population. Sci Rep. 2022 May 21;12(1):8622. doi: 10.1038/s41598-022-11787-4. PMID 35597776
- [Result] Robineau O, Wiernik E, Lemogne C, de Lamballerie X, Ninove L, Blanche H, Deleuze JF, Ribet C, Kab S, Goldberg M, Severi G, Touvier M, Zins M, Carrat F. Persistent symptoms after the first wave of COVID-19 in relation to SARS-CoV-2 serology and experience of acute symptoms: A nested survey in a population-based cohort. Lancet Reg Health Eur. 2022 Jun;17:100363. doi: 10.1016/j.lanepe.2022.100363. Epub 2022 Apr 12. PMID 35434687
- [Result] Carrat F, Lapidus N, Ninove L, Blanche H, Rahib D, Saba Villarroel PM, Touvier M, Severi G, Zins M, Deleuze JF, de Lamballerie X; SAPRIS-SERO study group. Age, COVID-19-like symptoms and SARS-CoV-2 seropositivity profiles after the first wave of the pandemic in France. Infection. 2022 Feb;50(1):257-262. doi: 10.1007/s15010-021-01731-5. Epub 2021 Nov 25. PMID 34822130
- [Result] Hoze N, Paireau J, Lapidus N, Tran Kiem C, Salje H, Severi G, Touvier M, Zins M, de Lamballerie X, Levy-Bruhl D, Carrat F, Cauchemez S. Monitoring the proportion of the population infected by SARS-CoV-2 using age-stratified hospitalisation and serological data: a modelling study. Lancet Public Health. 2021 Jun;6(6):e408-e415. doi: 10.1016/S2468-2667(21)00064-5. Epub 2021 Apr 8. PMID 33838700
- [Result] Lapidus N, Paireau J, Levy-Bruhl D, de Lamballerie X, Severi G, Touvier M, Zins M, Cauchemez S, Carrat F; SAPRIS-SERO study group. Do not neglect SARS-CoV-2 hospitalization and fatality risks in the middle-aged adult population. Infect Dis Now. 2021 Jun;51(4):380-382. doi: 10.1016/j.idnow.2020.12.007. Epub 2021 Jan 18. PMID 33521775
- [Result] Carrat F, de Lamballerie X, Rahib D, Blanche H, Lapidus N, Artaud F, Kab S, Renuy A, Szabo de Edelenyi F, Meyer L, Lydie N, Charles MA, Ancel PY, Jusot F, Rouquette A, Priet S, Saba Villarroel PM, Fourie T, Lusivika-Nzinga C, Nicol J, Legot S, Druesne-Pecollo N, Esseddik Y, Lai C, Gagliolo JM, Deleuze JF, Bajos N, Severi G, Touvier M, Zins M; for the SAPRIS and SAPRIS-SERO study groups. Antibody status and cumulative incidence of SARS-CoV-2 infection among adults in three regions of France following the first lockdown and associated risk factors: a multicohort study. Int J Epidemiol. 2021 Nov 10;50(5):1458-1472. doi: 10.1093/ije/dyab110. PMID 34293141
- [Result] Glemain B, Assaad C, Ghosn W, Moulaire P, de Lamballerie X, Zins M, Severi G, Touvier M, Deleuze JF; SAPRIS-SERO study group; Lapidus N, Carrat F, Ancel PY, Charles MA, Severi G, Touvier M, Zins M, Kab S, Renuy A, Le-Got S, Ribet C, Pellicer M, Wiernik E, Goldberg M, Artaud F, Gerbouin-Rerolle P, Enguix M, Laplanche C, Gomes-Rima R, Hoang L, Correia E, Barry AA, Senina N, Allegre J, Szabo de Edelenyi F, Druesne-Pecollo N, Esseddik Y, Hercberg S, Deschasaux M, Charles MA, Benhammou V, Ritmi A, Marchand L, Zaros C, Lordmi E, Candea A, de Visme S, Simeon T, Thierry X, Geay B, Dufourg MN, Milcent K, Rahib D, Lydie N, Lusivika-Nzinga C, Pannetier G, Lapidus N, Goderel I, Dorival C, Nicol J, Robineau O, Lai C, Belhadji L, Esperou H, Couffin-Cadiergues S, Gagliolo JM, Blanche H, Sebaoun JM, Beaudoin JC, Gressin L, Morel V, Ouili O, Deleuze JF, Ninove L, Priet S, Villarroel PMS, Fourie T, Mohamed Ali S, Amroun A, Seston M, Ayhan N, Pastorino B, de Lamballerie X. Revisiting the link between COVID-19 incidence and infection fatality rate during the first pandemic wave. Sci Rep. 2025 May 5;15(1):15638. doi: 10.1038/s41598-025-99078-6. PMID 40325150
- [Result] Pignon B, Wiernik E, Ranque B, Robineau O, Carrat F, Severi G, Touvier M, Gouraud C, Ouazana Vedrines C, Pitron V, Hoertel N, Kab S, Tebeka S, Goldberg M, Zins M, Lemogne C. SARS-CoV-2 infection and the risk of depressive symptoms: a retrospective longitudinal study from the population-based CONSTANCES cohort. Psychol Med. 2024 Oct 14;54(14):1-10. doi: 10.1017/S0033291724002435. Online ahead of print. PMID 39399920
- [Result] Glemain B, de Lamballerie X, Zins M, Severi G, Touvier M, Deleuze JF; SAPRIS-SERO study group; Lapidus N, Carrat F. Estimating SARS-CoV-2 infection probabilities with serological data and a Bayesian mixture model. Sci Rep. 2024 Apr 25;14(1):9503. doi: 10.1038/s41598-024-60060-3. PMID 38664455
- [Result] Charles MA, Ancel PY, Simeon T, Marchand-Martin L, Zaros C, Dufourg MN, Benhamou V, Blanche H, Deleuze JF, Rahib D, Lydie N, de Lamballerie X, Carrat F. SARS-CoV-2 seroprevalence in French 9-year-old children and their parents after the first lockdown in 2020. Front Pediatr. 2023 Oct 25;11:1274113. doi: 10.3389/fped.2023.1274113. eCollection 2023. PMID 37954429
- [Result] Ramillon J, de Lamballerie X, Robineau O, Blanche H, Severi G, Touvier M, Zins M, Carrat F; SAPRIS-SERO study group; SAPRIS study group; Lapidus N. Correction: Antibody response, associated symptoms and profile of patients presumably infected by SARS-CoV-2 with taste or smell disorders in the SAPRIS multicohort study. BMC Infect Dis. 2023 Jul 26;23(1):492. doi: 10.1186/s12879-023-08450-2. No abstract available. PMID 37495960
- [Result] Deschasaux-Tanguy M, Szabo de Edelenyi F, Druesne-Pecollo N, Esseddik Y, Allegre J, Srour B, Galan P, Hercberg S, Severi G, Zins M, Wiernik E; SAPRIS-SERO study group; de Lamballerie X, Carrat F, Touvier M. ABO blood types and SARS-CoV-2 infection assessed using seroprevalence data in a large population-based sample: the SAPRIS-SERO multi-cohort study. Sci Rep. 2023 Mar 23;13(1):4775. doi: 10.1038/s41598-023-30714-9. PMID 36959255